CLINICAL TRIAL: NCT01363986
Title: A Multicenter, Open Label Study to Assess the Effect of Trastuzumab + Whole Brain Radiotherapy (WBRT) on Brain Metastases From HER-2 Positive Breast Cancer. (bHERt-2)
Brief Title: A Study of Herceptin (Trastuzumab) in Combination With Whole Brain Radiotherapy in Patients With HER-2 Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was prematurely terminated due to difficulties experienced in recruiting patients in a reasonable timeframe.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25432
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (1):
- Trastuzumab Monotherapy (Experimental): Participants received an initial loading dose of 4 milligrams per kilogram (mg/kg) trastuzumab intravenous (i.v.), followed by weekly doses of 2 mg/kg i.v. for up to 18 weeks.
  Interventions: Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: trastuzumab [Herceptin] — Initial loading dose of 4 mg/kg i.v. infusion, followed by weekly doses of 2 mg/kg for up to 18 weeks.

SUMMARY:
This single-arm, multicenter, open-label study will evaluate the efficacy and safety of Herceptin (trastuzumab) in combination with whole brain radiotherapy on brain metastases in patients with HER-2 positive breast cancer. The patients will receive Herceptin 4 mg/kg (loading dose) followed by 2 mg/kg for a maximum of 18 weekly cycles. The anticipated time on study treatment is 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of breast carcinoma with HER-2 overexpression
* At least one measurable brain metastasis
* Patients for whom, according to investigator assessment, whole brain radiotherapy is the best therapeutic option
* Performance status (WHO) </=2
* Life expectancy >/=3 months

Exclusion Criteria:

* Presence of neoplastic meningitis
* Any prior radiotherapy to the brain
* Patients for whom, according to investigator assessment, stereotactic radiotherapy is the best therapeutic option
* Previous neoplasms, other than breast carcinoma, within 5 years since enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Italy (16):
  - Ancona
  - Brindisi
  - Candiolo
  - Florence
  - Latina
  - Lecce
  - Meldola
  - Parma
  - Ravenna
  - Roma
  - Rozzano
  - San Giovanni Rotondo
  - Saronno
  - Sassari
  - Torino
  - Viterbo

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab Monotherapy: Participants received an initial loading dose of 4 milligrams per kilogram (mg/kg) trastuzumab intravenously (i.v.) on Day 1, followed by doses of 2 mg/kg trastuzumab i.v. once weekly for up to 18 weeks.
Period: Overall Study
Arm/Group | Trastuzumab Monotherapy
Started | 3
Completed | 2
Not Completed | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all consented participants who received study treatment.
Groups:
- Trastuzumab Monotherapy: Participants received an initial loading dose of 4 mg/kg trastuzumab i.v. on Day 1, followed by doses of 2 mg/kg trastuzumab i.v. once weekly for up to 18 weeks.
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Brain Objective Response According to Response Evaluation Criteria In Solid Tumors (RECIST) Criteria at Cycle 7
Description: Brain objective response was defined as either a complete response (CR) or partial response (PR), provided that there was no increase in steroid requirements or worsening of neurological signs and symptoms. CR was defined as the disappearance of all central nervous system (CNS) lesions. PR was defined as a greater than or equal to (≥) 30 percent (%) reduction in the volumetric sum of all measurable CNS lesions.
Time Frame: Baseline and Cycle 7 (Week 7, approximately 5 weeks after completion of whole brain radiotherapy [WBRT])
Population: ITT population; 1 participant was not assessed at Cycle 7.
Measure: Number; unit: participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Number of Participants With Brain Objective Response According to RECIST Criteria at Cycle 15
Description: Brain objective response was defined as either a CR or PR, provided that there was no increase in steroid requirements or worsening of neurological signs and symptoms. CR was defined as the disappearance of all CNS lesions. PR was defined as ≥30% reduction in the volumetric sum of all measurable CNS lesions.
Time Frame: Baseline and Cycle 15 (Week 15, approximately 13 weeks after completion of WBRT)
Population: ITT population; 2 participants were not assessed at Cycle 15.
Measure: Number; unit: participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 1
participants | 0

3. Secondary Outcome: Number of Participants With Brain Objective Response Defined According to RECIST Criteria at the Final Visit
Description: Brain objective response was defined as either a CR or PR), provided that there was no increase in steroid requirements, or worsening of neurological signs and symptoms. CR was defined as the disappearance of all CNS lesions. PR was defined as ≥30% reduction in the volumetric sum of all measurable CNS lesions.
Time Frame: BL and 4 weeks after Cycle 15 (Week 15, approximately 13 weeks after completion of WBRT) or the last dose of study treatment
Population: ITT population; 1 participant was not assessed at the final visit.
Measure: Number; unit: participant
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 2
participant | 1

4. Secondary Outcome: Overall Survival
Description: The number of participants surviving at the final visit.
Time Frame: Baseline, weekly for 3 weeks (pre-WBRT phase), Cycles 1 through 15 (treatment phase Weeks 1 through 15), and 4 weeks after Cycle 15 (Week 15) or the last dose of study treatment
Population: ITT population; survival status of 1 participant was unknown at the final visit.
Measure: Number; unit: participant
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 2
participant | 1

5. Secondary Outcome: Brain Progression-Free Survival (B-PFS)
Description: B-PFS was defined as the time from the date of first study drug assumption and the date of documented evidence of brain progression (defined as appearance of new brain metastases or progression of pre-existing lesions) or death for brain progression, whichever came first. Progression in other metastatic sites, deaths not due to brain-progression and withdrawals due to adverse events were to be considered as competing risk.
Time Frame: as for outcome 4
Population: Due to the premature interruption of the study and the small number of enrolled participants (3 nerolled), all participant data were listed only, without any descriptive statistics or data analysis. The endpoint of B-PFS was thus not analyzed.
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from randomization up through 28 days after the final study drug treatment.
Description: Safety was assessed in all consented participants who received study treatment.
Arm/Group | Trastuzumab Monotherapy
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Monotherapy (N=3)
Nausea (Gastrointestinal disorders) | 1
Headache (General disorders) | 2
Asthenia (General disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 1
Epilepsy (Nervous system disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Device-related infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1
Speech disorder (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.